CLINICAL TRIAL: NCT05184764
Title: Phase 1b/2a, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of Safety, Tolerability, and Efficacy of Intravenous AP-SA02 as an Adjunct to Best Available Antibiotic Therapy for the Treatment of Adults With Bacteremia Due to Staphylococcus Aureus
Brief Title: Study Evaluating Safety, Tolerability, and Efficacy of Intravenous AP-SA02 in Subjects With S. Aureus Bacteremia
Acronym: diSArm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-SA02-101
Record Dates: First submitted 2021-11-24; First posted 2022-01-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-11

CONDITIONS: Bacteremia; Staphylococcus Aureus; Staphylococcus Aureus Bacteremia; Bacteremia Staph; Bacteremia Due to Staphylococcus Aureus
Keywords: Bacteriophage; Phage; Bacteremia; Staphylococcus Aureus; Staphylococcus; SAB
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AP-SA02 (Experimental): Anti-staphylococcal bacteriophage
  Interventions: Biological: AP-SA02
- Placebo (Placebo Comparator): Inactive isotonic solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AP-SA02 — Bacteriophage administered via intravenous bolus infusion
  Arms: AP-SA02
Other: Placebo — Inactive Placebo administered via intravenous bolus infusion
  Arms: Placebo

SUMMARY:
Phase 1b/2a, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Escalation Study of the Safety, Tolerability, and Efficacy of Intravenous AP SA02 as an Adjunct to Best Available Antibiotic Therapy Compared to Best Available Antibiotic Therapy Alone for the Treatment of Adults With Bacteremia Due to Staphylococcus aureus

DETAILED DESCRIPTION:
This study will be conducted in two phases: Phase 1b will to evaluate the safety and tolerability of multiple ascending intravenous (IV) doses of AP-SA02 or placebo as an adjunct to best available therapy (BAT) compared to BAT alone in subjects with SA bacteremia (SAB). Phase 2a will evaluate the efficacy, safety, and tolerability of multiple doses of AP-SA02 or placebo as an adjunct to BAT compared to BAT alone in subjects with complicated SAB.

ELIGIBILITY:
Key Inclusion Criteria:

* A hospitalized female or male ≥ 18 years old
* Positive blood culture for Staphylococcus aureus (SA)
* Source of SA infection controlled, or a plan for source control, if relevant
* Not pregnant or breastfeeding and is not of reproductive potential or agrees to use contraception if or reproductive potential

Key Exclusion Criteria:

* Concomitant growth of organisms besides SA
* Left-sided infectious endocarditis by modified Duke criteria
* Known or suspected brain abscess or meningitis
* Known allergy to phage products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (Safety and Tolerability) of multiple doses of intravenous AP-SA02 | Day 1 first dose through Day 12 or through End of Study for serious AEs
  Incidence and severity of treatment-emergent adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Clinical Improvement or Response at Day 12 | Day 12
  Description of clinical outcome in the Microbiological Intent-to-Treat (mITT) Population. Clinical outcome of improvement or response is defined as survival with resolution of S. aureus-related clinical signs and symptoms as well as eradication of S. aureus bacteremia, and without new foci of infection or complications of S. aureus bacteremia
Clinical Improvement or Response at 7 days after completion of antibiotic therapy | 7 days post completion of best available antibiotic therapy
  Description of clinical outcome in the Microbiological Intent-to-Treat (mITT) Population. Clinical outcome of improvement or response is defined as survival with resolution of S. aureus-related clinical signs and symptoms as well as eradication of S. aureus bacteremia, and without new foci of infection or complications of S. aureus bacteremia
Clinical Improvement or Response at End of Study | 28 days post completion of best available antibiotic therapy
  Description of clinical outcome in the Microbiological Intent-to-Treat (mITT) Population. Clinical outcome of improvement or response is defined as survival with resolution of S. aureus-related clinical signs and symptoms as well as eradication of S. aureus bacteremia, and without new foci of infection or complications of S. aureus bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Birx, MD, Study Director — Armata Pharmaceuticals, Inc.
Locations (28):
- United States (23):
  - Banner University Medical Center, Tucson, Arizona
  - University of California, San Diego (UCSD) - Medical Center, La Jolla, California
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - University of Florida (UF) - Division of Infectious Disease, Gainesville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - The Jamaica Hospital Medical Center, Jamaica, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina - Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Regional One Healthcare, Memphis, Tennessee
  - Methodist Hospital Research Institute - Houston, Houston, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Adelaide Hospital, Adelaide
  - Monash Health, Clayton
  - Royal Melbourne Hospital, Melbourne
  - The Alfred Hospital, Melbourne
  - Westmead Hospital, Westmead

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Armata Pharmaceuticals, Inc. — http://armatapharma.com